CLINICAL TRIAL: NCT04945174
Title: Stroke School - Cross-sectorial Physical Exercise for Patients With Minor Stroke or Non-disabling Stroke
Brief Title: Stroke School -Including Physical Exercise, Patient Education and Individual Follow-up Sessions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Christina Kruuse, Professor, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-20059985
Record Dates: First submitted 2021-04-27; First posted 2021-06-30 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-02

CONDITIONS: Minor Stroke; Non-disabling Stroke; Transient Ischemic Attack
Keywords: Minor stroke; Stroke prevention; Physical exercise; Patient education; Cardiorespiratory fitness; Non-disabling stroke
MeSH Terms: conditions — Ischemic Attack, Transient; Motor Activity | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Active Comparator): 12 weeks of supervised cardiorespiratory exercise twice a week (6 weeks at the hospital and 6 weeks in the local municipality) combined with patient education and individual follow-up sessions
  Interventions: Behavioral: Cardiorespiratory exercise combined with patient education and individual follow-up sessions
- Usual care (No Intervention): The usual care group is encouraged to perform home-based aerobic exercise on their own

INTERVENTIONS:
Behavioral: Cardiorespiratory exercise combined with patient education and individual follow-up sessions — 6 weeks of cardiorespiratory exercise combined with patient education at the hospital, followed by 6 weeks of cardiorespiratory exercise in the local municipality. Subsequently individual follow-up sessions with the aim to facilitate the patients to stay physically active in their everyday life
  Arms: Exercise

SUMMARY:
In a randomized controlled trial the effect of 12 weeks of cross-sectorial physical exercise combined with patient education and individual follow-up session is investigated in patients with minor stroke or non-disabling stroke.

DETAILED DESCRIPTION:
Hypertension and physical inactivity are the most common risk factors for stroke. Patients with minor stroke or transient ischemic attack (TIA) have short-lasting symptoms, often with remission within hours or days. Though patients experience a quick remission, they have an increased risk of a recurrent stroke and progressive cognitive dysfunction. The patients are also likely to have other disposing risk factors such as diabetes, smoking, and hypercholesterolemia which may increase the risk of a recurrent stroke. Following hospital discharge, the patients are offered preventive medication, but no standardized rehabilitation or exercise. Previous studies have shown that physical exercise decreases cardiovascular risk factors for patients after stroke and increases physical function and quality of life.

The aim is to develop and evaluate a standardized exercise program (a stroke school) for patients with minor stroke or TIA. The intervention consist of 6 weeks of supervised aerobic exercise at the hospital combined with patient education including knowledge on stroke risk factors. Subsequently, 6 weeks of supervised aerobic exercise in their local municipality. After the 12 weeks of exercise, patients are offered individual, motivational follow-up sessions with the purpose to facilitate the patients to stay physically active in their everyday life.

This intervention will increase the patients´ knowledge regarding risk factors for stroke and cardiovascular disease, increase their cardiorespiratory fitness and facilitate the patients to be physical active and hopefully slow the progression of vascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a minor stroke or TIA without the need of rehabilitation after hospital discharge, but need physical activity in order to prevent cardiovascular diseases
* Patients spending ≤ 5 hour of leisure time on high-intensity physical activity on weekly basis within the last 3 months
* Able to speak and read Danish and to provide informed consent
* Individuals ≥ 18 years of age

Exclusion Criteria:

* Previous large-artery stroke or hemorrhagic stroke
* Unstable cardiac condition, e.g. pacemaker
* Uncontrolled hypertension (patients not responding adequately to antihypertensive medication when applying treatment according to guidelines)
* Symptoms or comorbidities not allowing exercise on a stationary bicycle (e.g. claudication)
* Dyspnoea caused by heart or pulmonary disease (e.g. COPD)
* Aphasia, or dementia that interferer with understanding the protocol and/or physical examinations.
* Patients diagnosed with dementia at hospital admission (a score ≤23/30 on the Mini-Mental State Examination are not invited into the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Change in 'the Graded Cycling Test with Talk Test' from baseline to 3 months | from baseline to 3 months (post-intervention)
  A sub-maximal exercise test on a stationary bicycle where the workload increases by 15 Watts (W) every minute and each minute the patient recites a standardized text passage. When the patient is no longer able to speak comfortably the test terminates. The higher score the better cardiorespiratory fitness

SECONDARY OUTCOMES:
Change in Physical Activity Scale | from baseline to 3 months (post-intervention)
  A questionnaire measuring number of hours of self-reported physical activity during daily living. It reveals daily time spent on sleep, sitting down at work, standing/walking at work, heavy physical work during working hours, active commuting to/from work, and sedentary behavior, including television watching and reading. Additionally, the patients record the weekly time spent on light-intensity, moderate-intensity, and vigorous-intensity activity during leisure time.
Change in Physical Activity Scale from baseline to 12-months post-stroke | From baseline to 12-months post-stroke
  A questionnaire measuring number of hours of self-reported physical activity during daily living. It reveals daily time spent on sleep, sitting down at work, standing/walking at work, heavy physical work during working hours, active commuting to/from work, and sedentary behavior, including television watching and reading. Additionally, the patients record the weekly time spent on light-intensity, moderate-intensity, and vigorous-intensity activity during leisure time.
Change in maximum cardiopulmonary exercise test from baseline to 3 months post-stroke | from baseline to 3 months (post-intervention)
  A maximal exercise test on a stationary bicycle
Change in The WHO-5 Well-being index from baseline to to 3 months post-stroke | from baseline to 3 months (post-intervention)
  A questionnaire measuring current mental well-being on a scale from 0-100 points where higher points indicates better mental well-being
Change in The WHO-5 Well-being index from baseline to 12-months post-stroke | From baseline to 12-months post-stroke
  A questionnaire measuring current mental well-being on a scale from 0-100 points where higher points indicates better mental well-being
Change in Montreal Cognitive Assessment from baseline to 3 months post-stroke | from baseline to 3 months (post-intervention)
  A cognitive screening test for detection of mild cognitive impairments, the score ranges from 0-30 points and a high score indicates better cognitive function
Change in Montreal Cognitive Assessment from baseline to 12-months post-stroke | From baseline to 12-months post-stroke
  A cognitive screening test for detection of mild cognitive impairments, the score ranges from 0-30 points and a high score indicates better cognitive function
Change in Anxiety and depression from baseline to 3 months post-stroke | from baseline to 3 months (post-intervention)
  This is a self-reported questionnaire that measures anxiety and depression. A total score of 0-21 points is possible, with a higher score indicating more severe symptoms of depression or anxiety.
Change in Anxiety and depression from baseline 12-months post-stroke | From baseline 12-months post-stroke
  This is a self-reported questionnaire that measures anxiety and depression. A total score of 0-21 points is possible, with a higher score indicating more severe symptoms of depression or anxiety.
Change in Fatigue Severity Scale from baseline to 3 months post-stroke | from baseline to 3 months (post-intervention)
  A 20-item self-report instrument designed to measure fatigue. The score ranges from 9-63 points, and a higher score indicates greater severity of fatigue
Change in Fatigue Severity Scale from baseline to 12-months post-stroke | From baseline to 12-months post-stroke
  A 20-item self-report instrument designed to measure fatigue. The score ranges from 9-63 points, and a higher score indicates greater severity of fatigue
Change in The Multidimensional Fatigue Inventory from baseline to 3-months post-stroke | From baseline to 12-months post-stroke
  Four questions on General fatigue is calculated on a score from 4-20, with higher scores representing increased fatigue
Change in The Multidimensional Fatigue Inventory from baseline to 12-months post-stroke | From baseline to 12-months post-stroke
  Four questions on General fatigue is calculated on a score from 4-20, with higher scores representing increased fatigue
Change in blood pressure from baseline to 3 months post-stroke | from baseline to 3 months (post-intervention)
  Assessment of blood pressure (systolic and diastolic)
Change in blood pressure from baseline to 12-months post-stroke | From baseline to 12-months post-stroke
  Assessment of blood pressure (systolic and diastolic)
Change in body mass index from baseline to 3 months post-stroke | from baseline to 3 months (post-intervention)
  Measures of weight in kilograms, and height in meters will be aggregated to arrive at one reported value, the body mass index (kg/m^2).
Change in body mass index from baseline to 12-months post-stroke | From baseline to 12-months post-stroke
  Measures of weight in kilograms, and height in meters will be aggregated to arrive at one reported value, the body mass index (kg/m^2).
Change in Modified rankin scale from baseline to 3 months post-stroke | from baseline to 3 months (post-intervention)
  A measurement of symptoms/motor function. The score ranges from 0-6 points, where 0 represents "no symptoms at all" and 6 points represents "dead".
Change in Modified rankin scale from baseline to 12-months post-stroke | From baseline to 12-months post-stroke
  A measurement of symptoms/motor function. The score ranges from 0-6 points, where 0 represents "no symptoms at all" and 6 points represents "dead".
Change in high-sensitivity C-reactive protein from baseline to 3 months post-stroke | from baseline to 3 months (post-intervention)
  Blood samples to evaluate degree of inflammation (low risk: < 1 mg/L, average risk: 1-3 mg/L, and high risk: >3 mg/L).
Change in high-sensitivity C-reactive protein from baseline to 12-months post-stroke | From baseline to 12-months post-stroke
  Blood samples to evaluate degree of inflammation (low risk: < 1 mg/L, average risk: 1-3 mg/L, and high risk: >3 mg/L).
Change in Pro brain natriuretic peptid from baseline to 3 months post-stroke | from baseline to 3 months (post-intervention)
  Blood samples to evaluate cardiac function (normal: < 125 pg/mL, critical value: > 400 pg/mL)
Change in Pro brain natriuretic peptid from baseline to 12-months post-stroke | From baseline to 12-months post-stroke
  Blood samples to evaluate cardiac function (normal: < 125 pg/mL, critical value: > 400 pg/mL)
Change in Cathepsin B from baseline to 3 months post-stroke | from baseline to 3 months (post-intervention)
  Blood samples to evaluate muscle protein. (high level of Cathepsin B may associate to improve cognitive function)
Change in Cathepsin B from baseline to 12-months post-stroke | From baseline to 12-months post-stroke
  Blood samples to evaluate muscle protein. (high level of Cathepsin B may associate to improve cognitive function)
Change in Magnetic Resonance Imaging from baseline to 12-months post-stroke | From baseline to 12-months post-stroke
  detection of number of new infarcts or white matter lesions
Change in the Stages of exercise behavior change from baseline to 3 months post-stroke | from baseline to 3 months (post-intervention)
  A questionnaire consisting of six categories describing differerent stages towards exercise behavior change, ranking from no intention to change behavior (precontemplation) to sustain behavior change (maintenance).
  Data will be analysed by calculating the number of patients (percentage) in each category and with a comparison between groups
Change in the Stages of exercise behavior change from baseline to 12-months post-stroke | From baseline to 12-months post-stroke
  A questionnaire consisting of six categories describing differerent stages towards exercise behavior change, ranking from no intention to change behavior (precontemplation) to sustain behavior change (maintenance).
  Data will be analysed by calculating the number of patients (percentage) in each category and with a comparison between groups

OTHER OUTCOMES:
Number of patients with cardiovascular event from baseline to 5 years post-stroke | 5 years post-stroke
  Follow-up 5 years from inclusion on cardiovascular events
Number of patients who have died from baseline to 5 years post-stroke | 5 years post stroke
  Follow-up 5 years from inclusion on death

CONTACTS AND LOCATIONS:
Overall Officials: Christina Kruuse, Professor, Principal Investigator — Herlev Gentofte Hospital, Department of Neurology; Anders Hougaard, MD, Ph.d., Study Director — Herlev Gentofte hospital, Department of Neurology,
Locations (2):
- Denmark (2):
  - Herlev Hospital, Copenhagen, Herlev
  - Department of Neurology, Herlev-Gentofte Hospital, Herlev

IPD SHARING:
Plan to Share IPD: No